CLINICAL TRIAL: NCT03948516
Title: Validation of a Point-of-care Screening Tool for Children With Sickle Cell Disease
Brief Title: Sickle Cell Disease, Hemechip
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: US federal government (Unknown); University of Nebraska (Other); University of North Carolina, Chapel Hill (Other); Case Western Reserve University (Other); Aminu Kano Teaching Hospital, Nigeria (Unknown); Murtala Muhammad Specialist Hospital, Nigeria (Unknown); Hasiya Bayero Hospital, Nigeria (Unknown)
Responsible Party: Principal Investigator, AOwusu-Ansah, Physician, University Hospitals Cleveland Medical Center
Other Study IDs: 04-17-15
Record Dates: First submitted 2019-05-01; First posted 2019-05-14 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants tested for Sickle cell disease

SUMMARY:
Sickle cell disease is very common in Nigeria. Early diagnosis is important to prevent or reduce serious complications from the disease and to enable children stay healthy. To this end, the investigators would like to test a new, simple and quick device called the HemeChip to determine if it can detect whether or not someone has sickle cell disease. The investigators will compare the results obtained with the HemeChip with a standard method of diagnosing sickle cell disease known as Isoelectric focusing (IEF) or High Performance Liquid Chromatography (HPLC).If the investigators show that the new device can differentiate between children who have sickle cell disease and those who don't as successfully as the IEF or HPLC, they estimate a sharp increase in the use of this device in many countries especially in Africa due to its lower cost

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a group of inherited disorders of haemoglobin (Hb) synthesis, first described in the medical literature by James Herrick in 1910. Each year about 300,000 infants are born with SCD, including more than 200,000 cases in subSaharan Africa alone. In Nigeria alone, there are over 150,000 of these children born annually and it is estimated that between 50-90% of these children die before their fifth birthday. Overall, in the region, 6% of all childhood mortality in children less than 5 years of age is due to SCD complications and infections. Vaso occlusive crisis and anemia are serious complications of SCD, with infection often being the major cause of hospitalizations, crisis and death. SCD is caused by a point mutation in the sixth codon of the beta globin chain that produces normal Hb (HbA). This substitution of hydrophilic glutamic acid with hydrophobic valine produces sickle Hb (HbS), which is abnormally polymerized at low oxygen conditions causing sickling. Abnormal polymerization of HbS affects red cell membrane properties, shape, and density, and subsequent critical changes in inflammatory cell and endothelial cell function.

The clinical consequences of SCD include painful crises, widespread organ damage, and early mortality. Current standard practices for diagnosing SCD are high performance liquid chromatography (HPLC) and bench-top Hb electrophoresis. These two approaches, however, require trained personnel and state-of-the-art facilities, both of which may be lacking in many parts of sub-Saharan Africa where the disease is most prevalent.

These laboratory methods also carry significant costs which may be unaffordable for most patients. HemeChip diagnostic system offers an original and innovative solution, leveraging a novel engineering approach, to point of care (POC) diagnosis of SCD. HemeChip separates haemoglobin protein types in a miniscule volume of blood (1μL) on a piece of cellulose acetate paper that is housed in a micro-engineered chip with a controlled environment and electric field. Differences in Hb mobilities allow separation to occur within the cellulose acetate paper. A micro-engineered design and multiple layer lamination approach are utilized in fabricating the HemeChip. The design allows rapid manual assembly and results are available within a few minutes of performing the test.

HemeChip can also integrate with a mobile user interface (e.g. IPhone, IPod), which shows the test result quantitatively and objectively on the screen. HemeChip can be used by anyone after a short (30 minute) training, eliminating the need for highly skilled personnel.

ELIGIBILITY:
Inclusion Criteria:

* Fever or hypothermia (Temp ≥38 C or ≤36 C) Plus one of the following (prostration, excessive crying, poor feeding, altered consciousness, convulsion, difficulty breathing, profuse vomiting, diarrhea) & rapid breathing (0-2months>60 breaths/min, 3-12months >50 breaths/min, 13- 59 months > 40 breaths /min)
* Provision of signed and dated written informed consent by parent or guardian

Exclusion Criteria:

* Parent of child chooses to opt out of the study after initial consent.
* Blood transfusion within 3 months of study enrollment.
* Presence of condition or abnormality that in the opinion of the investigator would compromise the safety of the child or the quality of the data.

Ages: 6 Weeks to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants and children aged 6 weeks to 60 months
Sampling Method: Probability Sample
Enrollment: 738 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Validation of the HemeChip technology as a novel, point-of-care (POC) platform for screening SCD. | 30 minutes
  The results obtained using the HemeChip will be compared to High Performance Liquid Chromatography (HPLC), and the sensitivity and specificity of the HemeChip will be determined.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- Nigeria (3):
  - Aminu Kano Teaching Hospital, Kano
  - Hasiya Bayero Pediatric Hospital, Kano
  - Murtala Mohammed Specialist Hospital, Kano

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT03948516/Prot_SAP_000.pdf